CLINICAL TRIAL: NCT04383119
Title: A Randomized Phase II Trial Comparing the Activity of trabectedIn vs Gemcitabine in Patients With Metastatic or Locally Advanced Leiomyosarcoma Pretreated With Conventional Chemotherapy
Brief Title: Trial in Patients With Metastatic or Locally Advanced Leiomyosarcoma
Acronym: ISG-ARTICLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISG-ARTICLE
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Leiomyosarcoma of Ovary; Soft Tissue Sarcoma
Keywords: advanced leiomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, open-label, two arms with crossover. Patients will be randomized to receive Trabectedin (arm A) or Gemcitabine (arm B).
  In case of progressive disease (PD) or unacceptable toxicity during the assigned treatment, the patient will switched to the other arm
Masking Description: Not applicable (open label study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Trabectedin at the dose of 1.5 mg/m2-1.3 mg/m2 with a top-dose of 2.6 total mg per cycle (according the clinical practice in pretreated patients and in all our ISG studies) will be administered via a central venous catheter as a 24-hour infusion on day 1 of 21-days treatment cycles
  Interventions: Drug: Trabectedin
- Arm B (Active Comparator): Gemcitabine 800-1000 mg/m2 will be administered via a central venous catheter on days 1,8 every 21 days
  Interventions: Drug: Gemcitabine
- Observational Cohort (Active Comparator): Treatmen according clinical practice (not defined in advance). The patient who will refuse randomization between Arm A and B can choose to participate to the observational cohort to the study, where they will be treated according clinical practice
  Interventions: Drug: No Intervention: Observational Cohort

INTERVENTIONS:
Drug: Trabectedin — Trabectedin in monotherapy
  Other Names: Trabectedin arm
  Arms: Arm A
Drug: Gemcitabine — Gemcitabine, control arm
  Other Names: Gemcitabine arm
  Arms: Arm B
Drug: No Intervention: Observational Cohort — Treatment according clinical practice
  Arms: Observational Cohort

SUMMARY:
Study is aimed at evaluating the activity of Trabectedin (arm A) in advanced leiomyosarcomas, having Gemcitabine (arm B) as the comparator.

In addition to the randomized cohort, the study has also an observational prospective cohort which include patients who will refuse the randomization or for whom the investigator will not judge the randomization as an appropriate option.

In order to allow the participation of sites only to the prospective-observational (non randomized) cohort, it was introduced the possibility to participate to the study and receive the ethical approval only to the Observational Prospective Cohort In parallel an optional translational study will be performed, in both cohorts, to identify factors predictive of the activity of Trabectedin or Gemcitabine in this specific histotype.

DETAILED DESCRIPTION:
The management of patients with leiomyosarcomas determines many difficulties. Despite patients with metastatic disease at diagnosis or who recur after initial treatment have a dismal prognosis and, except for a subset of selected patients with completely resectable disease, the median survival is less than two years.

At the advanced-disease stage, the main aim of treatment is to improve patient's quality of life, possibly survival, with the best compromise between toxicity and symptoms. Trabectedin (T) is a marine-derived cytotoxic approved by European MEdicine Agency (EMEA) and FDA.

It is indicated for the treatment of patients with advanced soft tissue sarcoma, after failure of anthracyclines-based chemotherapy or who are unsuitable to receive these agents.

Among Soft Tissue Sarcoma (STS), activity has been mainly detected in synovial sarcoma, liposarcoma and leiomyosarcoma. Although the response rate did not exceed 10%, T was demonstrated to provide disease control, with progression arrest rates exceeding 50% and progression-free survival rates exceeding 20% at 6 months. So far no phase II or III studies have been addressed to test the activity of T in leiomyosarcoma specifically (without differentiation between site of primary localization) in comparison with Gemcitabine.

This study is aimed at evaluating the activity of Trabectedin (arm A) in advanced leiomyosarcomas, having Gemcitabine (arm B) as the comparator. In parallel an optional translational study will be performed to identify factors predictive of the activity of Trabectedin or Gemcitabine in this specific histotype.

In addition to the randomized cohort, the study has also an observational prospective cohort which include patients who will refuse the randomization or for whom the investigator will not judge the randomization as an appropriate option.

In order to allow the participation of sites only to the prospective-observational (non randomized) cohort, it was introduced the possibility to participate to the study and receive the ethical approval only to the Observational Prospective Cohort In parallel an optional translational study will be performed, in both cohorts, to identify factors predictive of the activity of Trabectedin or Gemcitabine in this specific histotype.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of leiomyosarcoma
2. Patients with diagnosis of unresectable or metastatic leiomyosarcoma
3. Patients who received at least on previous systemic treatment with anthracycline-based chemotherapy.
4. Patients suitable to receive gemcitabine or trabectedin therapy.
5. Measurable or evaluable disease with RECIST 1.1 criteria.
6. Evidence of progression according RECIST 1.1 during the 6 months before study entry.
7. Age ≥18 years
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
9. All previous anticancer treatments must have completed ≥ 3 weeks prior to first dose of study drug.
10. The patient has resolution of adverse events, with the exception of alopecia, and of all clinically significant toxic effects of prior loco-regional therapy, surgery, radiotherapy or systemic anticancer therapy to ≤ Grade 1, by National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
11. Adequate bone marrow, liver and renal function
12. Left Ventricular Ejection Fraction ≥ 50% and/or above lower institutional limit of normality.
13. Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation each cycle of chemotherapy.
14. No history of arterial and/or venous thromboembolic event within the previous 12 months.
15. The patient or legal representative must be able to read and understand the informed consent form and must have been willing to give written informed consent prior to any study specific procedure. The subject may also provide an optional consent for the biological/translational sub-study associated.

Exclusion Criteria:

1. Prior treatment with Trabectedin and/or Gemcitabine
2. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
3. History of other malignancies (except basal cell carcinoma or cervical carcinoma in situ, adequately treated), unless in remission from 5 years or more and judged of negligible potential of relapse.
4. Persistent toxicities with the exception of alopecia, caused by previous anticancer therapies
5. Metastatic brain or meningeal tumors
6. Active viral hepatitis
7. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus
8. Patients with any severe and/or uncontrolled medical conditions
9. Medical history of hemorrhage or a bleeding event ≥ Grade 3 (NCI-CTCAE v 5.0) within 4 weeks prior to the initiation of study treatment
10. Active clinically serious infections
11. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus
12. Previous treatment with radiation therapy within 14 days of first day of study drug dosing,
13. Major surgery within 4 weeks prior to study entry
14. Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors
15. Concomitant use of known strong or moderate CYP3A inducers
16. Patients undergoing renal dialysis or with Creatinin Clearance <30 ml/min or Creatinine >1,5 mg/dL
17. Pregnant or breast feeding patients
18. Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the Growth Modulation Index (GMI) in patients treated with Trabectedin or Gemcitabine in second line | Week 6, week 12, week 18, week 27, week 36 and week 45
  Ratio of Time To Progression with the nth line (TTPn) of therapy to the TTPn-1 with the n-1th line.

SECONDARY OUTCOMES:
Overall Response Rate | Week 6, week 12, week 18, week 27, week 36 and week 45
  Overall response rate according Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Overall Survival (OS) | 3 years and 5 years
  Survival from the first dose treatment to death for any cause
Progression free Survival (PFS) | 6 months
  Survival without disease progression
Duration of response | Week 6, week 12, week 18, week 27, week 36 and week 45
  Duration of tumor control according Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Adverse events related to the treatment | Week 3, week 6, week 9, week 12, week 18, week 27, week 36, week 45
  Safety in term of adverse event is evaluate from the first treatment dose throughout the study according to CTCAE 5.0
Compare the Growth Modulation Index (GMI) in patients treated with Trabectedin or Gemcitabine after second line | Week 6, week 12, week 18, week 27, week 36 and week 45
  Ratio of Time To Progression with the Mth line (TTPn) of therapy to the TTPn-1 with the n-1th line.

OTHER OUTCOMES:
Exploratory objectives | week 6, and at up to week 53
  Identify gene mutations that may be associated to response/resistance to the treatment and to clinical outcomes parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vincenzi, Prof/MD, Principal Investigator — Campus Biomedico of Rome
Locations (17):
- Italy (17):
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna, BO
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola, FC
  - Nuovo Ospedale di Prato, Prato, Firenze
  - Istituto Clinico Humanitas, Rozzano, MI
  - Centro di Riferimento Oncologico di Aviano, Aviano, PD
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - IRCCS Fondazione Piemonte per l'Oncologia, Candiolo, Torino
  - A.O.U.San Luigi Gonzaga, Orbassano, Torino
  - Istituto Ortopedico Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - H.San Martino di Genova, Genova
  - Fondazione IRCCS INT Milano, Milan
  - Istituto Europeo di Oncologia, Milan
  - IRCCS Istituto nazionale Tumori "Fondazione G.Pascale", Napoli
  - Irccs Istituto Oncologico Veneto (Iov), Padua
  - Ospedale Giaccone, Palermo
  - Istituto Regina Elena - IFO, Rome
  - ASL Città di Torino (Dipartimento di Oncologia), Torino

IPD SHARING:
Plan to Share IPD: No
Not applicable no plan to share IPD

REFERENCES:
- [Background] Hensley ML, Miller A, O'Malley DM, Mannel RS, Behbakht K, Bakkum-Gamez JN, Michael H. Randomized phase III trial of gemcitabine plus docetaxel plus bevacizumab or placebo as first-line treatment for metastatic uterine leiomyosarcoma: an NRG Oncology/Gynecologic Oncology Group study. J Clin Oncol. 2015 Apr 1;33(10):1180-5. doi: 10.1200/JCO.2014.58.3781. Epub 2015 Feb 23. PMID 25713428
- [Background] Pautier P, Floquet A, Chevreau C, Penel N, Guillemet C, Delcambre C, Cupissol D, Selle F, Isambert N, Piperno-Neumann S, Thyss A, Bertucci F, Bompas E, Alexandre J, Collard O, Lavau-Denes S, Soulie P, Toulmonde M, Le Cesne A, Lacas B, Duffaud F; French Sarcoma Group. Trabectedin in combination with doxorubicin for first-line treatment of advanced uterine or soft-tissue leiomyosarcoma (LMS-02): a non-randomised, multicentre, phase 2 trial. Lancet Oncol. 2015 Apr;16(4):457-64. doi: 10.1016/S1470-2045(15)70070-7. Epub 2015 Mar 18. PMID 25795402
- [Background] Demetri GD, Chawla SP, von Mehren M, Ritch P, Baker LH, Blay JY, Hande KR, Keohan ML, Samuels BL, Schuetze S, Lebedinsky C, Elsayed YA, Izquierdo MA, Gomez J, Park YC, Le Cesne A. Efficacy and safety of trabectedin in patients with advanced or metastatic liposarcoma or leiomyosarcoma after failure of prior anthracyclines and ifosfamide: results of a randomized phase II study of two different schedules. J Clin Oncol. 2009 Sep 1;27(25):4188-96. doi: 10.1200/JCO.2008.21.0088. Epub 2009 Aug 3. PMID 19652065
- [Background] Patel SR, Gandhi V, Jenkins J, Papadopolous N, Burgess MA, Plager C, Plunkett W, Benjamin RS. Phase II clinical investigation of gemcitabine in advanced soft tissue sarcomas and window evaluation of dose rate on gemcitabine triphosphate accumulation. J Clin Oncol. 2001 Aug 1;19(15):3483-9. doi: 10.1200/JCO.2001.19.15.3483. PMID 11481354
- [Background] Pautier P, Floquet A, Penel N, Piperno-Neumann S, Isambert N, Rey A, Bompas E, Cioffi A, Delcambre C, Cupissol D, Collin F, Blay JY, Jimenez M, Duffaud F. Randomized multicenter and stratified phase II study of gemcitabine alone versus gemcitabine and docetaxel in patients with metastatic or relapsed leiomyosarcomas: a Federation Nationale des Centres de Lutte Contre le Cancer (FNCLCC) French Sarcoma Group Study (TAXOGEM study). Oncologist. 2012;17(9):1213-20. doi: 10.1634/theoncologist.2011-0467. Epub 2012 Aug 20. PMID 22907974
- [Background] Seddon B, Strauss SJ, Whelan J, Leahy M, Woll PJ, Cowie F, Rothermundt C, Wood Z, Benson C, Ali N, Marples M, Veal GJ, Jamieson D, Kuver K, Tirabosco R, Forsyth S, Nash S, Dehbi HM, Beare S. Gemcitabine and docetaxel versus doxorubicin as first-line treatment in previously untreated advanced unresectable or metastatic soft-tissue sarcomas (GeDDiS): a randomised controlled phase 3 trial. Lancet Oncol. 2017 Oct;18(10):1397-1410. doi: 10.1016/S1470-2045(17)30622-8. Epub 2017 Sep 4. PMID 28882536